CLINICAL TRIAL: NCT07025148
Title: Switching From Clopidogrel to Low-dose Prasugrel in Patients at Dual-risk Following Percutaneous Coronary Intervention (TAILOR-BLEED-2)
Brief Title: Dual Antiplatelet Therapy Escalation From Standard-dose Clopidogrel to Low-Dose Prasugrel in Patients With High Bleeding and Ischemic Risk Undergoing PCI: A Prospective, Randomized Pharmacodynamic Study (TAILOR-BLEED-2)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202401774
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Coronary Arterial Disease (CAD); Percutaneous Coronary Intervention (PCI)
Keywords: Coronary artery disease; Dual antiplatelet therapy; High bleeding risk
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dual risk - Clopidogrel-based DAPT (Experimental): Patients deemed at high risk for both bleeding and ischemic risk randomized to continue clopdiogrel-based DAPT. High bleeding riks will be defined according to the Academic Research Consortium definition, while high ischemic risk will be defined as those patients with an ABCD-GENE score of 10 or higher.
  Interventions: Drug: Clopidogrel
- Dual risk - Low-dose prasugrel-based DAPT (Experimental): Patients deemed at high risk for both bleeding and ischemic risk randomized to receive low-dose prasugrel-based DAPT. High bleeding riks will be defined according to the Academic Research Consortium definition, while high ischemic risk will be defined as those patients with an ABCD-GENE score of 10 or higher.
  Interventions: Drug: Prasugrel
- Control (Active Comparator): Patients deemed at high risk for both bleeding but not at high risk for ischemic events being actively treated with clopidogrel-based DAPT as per standard of care. High bleeding riks will be defined according to the Academic Research Consortium definition.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 5 mg od for 30 ± 5 days
  Arms: Dual risk - Low-dose prasugrel-based DAPT
Drug: Clopidogrel — Clopidogrel 75 mg od for 30 ± 5 days
  Arms: Control; Dual risk - Clopidogrel-based DAPT

SUMMARY:
The primary aim of this study is to investigate the PD effects of switching from standard-dose clopidogrel dose to low-dose prasugrel versus continuing standard-dose clopidogrel in patients at dual-risk (HBR defined as the HBR-ARC criteria and HIR defined as ABCD-GENE score ≥10) following PCI. We hypothesize that in patients at dual-risk, switching from standard-dose clopidogrel to low-dose prasugrel will be superior to continuing standard-dose clopidogrel in terms of platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high bleeding risk (defined according to the ARC-HBR criteria) who have undergone PCI and are on maintenance treatment with DAPT, consisting of low-dose aspirin (81mg qd) with clopidogrel (75 mg qd) as part of standard of care for at least 30 days.
* Age ≥18 years.
* Provide written informed consent.

Exclusion Criteria:

* Prior cerebrovascular event.
* PCI within 30 days.
* Hemodynamic instability.
* On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban) or chronic low-molecular-weight heparin (at venous thrombosis treatment, not for prophylaxis).
* Hypersensitivity to Aspirin, Clopidogrel, or Prasugrel.
* Known hematologic malignancies or thrombocytopenia (platelet count <80x106/mL).
* Known hemoglobinopathies or anemia (hemoglobin <9 g/dL)
* Pregnant and breastfeeding women [women of childbearing age must use reliable birth control (i.e., oral contraceptives) while participating in the study].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity measured as PRU | 30 Day
  The primary end point of our study will be levels of platelet reactivity, measured as P2Y12 reaction units (PRU) using the VerifyNow system in patients at dual-risk (both HBR and HIR [ABCD-GENE score ≥10 points]) between low-dose prasugrel (5 mg qd) vs. standard-dose clopidogrel (75 mg qd)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Study Chair — University of Florida College of Medicine - Jacksonville; Luis Ortega-Paz, MD, PhD, Principal Investigator — University of Florida College of Medicine - Jacksonville
Locations (1):
- University of Florida Health, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared upon reasonable request to the primary investigator.
Supporting Information: Study Protocol
Time Frame: Individual patient data will be shared upon reasonable request to the primary investigator after publication of the primary results.
Access Criteria: Individual patient data will be shared upon reasonable request to the primary investigator.